CLINICAL TRIAL: NCT00060450
Title: Inhaled Nitric Oxide in Prevention/Treatment of Ischemia-Reperfusion Lung Injury Related to Lung Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MACIN1
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Ischemia-Reperfusion Injury
Keywords: Ischemia-reperfusion lung injury; IRLI
MeSH Terms: conditions — Reperfusion Injury | interventions — Nitric Oxide; Inhalation; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Inhaled Nitric Oxide
  Interventions: Drug: nitric oxide for inhalation
- 2 (Placebo Comparator): Placebo gas
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nitric oxide for inhalation — Either 10 or 20 ppm of inhaled nitric oxide for 24 hour post transplant
  Other Names: INOmax®
  Arms: 1
Drug: Placebo — Placebo gas will be given at 10 or 20 ppm for 24 hours post transplant
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effects of inhaled nitric oxide on both short-term physiology as well as on the development of ischemia-reperfusion lung injury (IRLI) in the immediate post transplant period. The specific hypothesis is that inhaled NO post lung transplantation will improve gas exchange/hemodynamic and thus reduce the development of post transplant IRLI.

DETAILED DESCRIPTION:
The objective is to determine the role of inhaled NO in the prevention/treatment of IRLI in lung transplant patients. The plan is to accomplish this objective in 2 phases:

Phase 1 - patients immediately post transplant will have a variety of physiologic measurements performed while breathing 0, 10, and 20 ppm inhaled NO. For the next 24 hours they will be kept on a mixture providing the best oxygen delivery and pulmonary artery pressure. Our specific aims in this phase are to characterize physiologic responses to inhaled NO and determine the incidence of IRLI in these patients over 24 hours.

Phase 2 - patients immediately post transplant will be randomized to either INO or placebo gas and followed for 24 hours. Our specific aim in this phase is to compare the rate of development of IRLI in the two groups.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing lung transplantation

Exclusion criteria:

* Participation in other experimental protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
arterial and mixed venous blood gases | first 4 hours post transplant
pulmonary vascular pressures | first 4 hours post transplant

SECONDARY OUTCOMES:
cardiac output | first 4 hours post transplant
systemic hemodynamics | first 4 hours post transplant
NO2 and NO concentrations | duration of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacIntyre, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States